CLINICAL TRIAL: NCT06528821
Title: Artificial Intelligence-Powered Electrocardiogram Detecting Culprit Vessel Blood Flow Abnormality in Acute Coronary Syndromes
Brief Title: AI-Powered ECG Detecting Culprit Vessel Blood Flow Abnormality in ACS
Acronym: AI-ECG-TIMI
Status: Recruiting | Type: Observational
Sponsor: Powerful Medical (Other)
Responsible Party: Sponsor
Other Study IDs: AI-ECG-TIMI_v1
Record Dates: First submitted 2024-07-26; First posted 2024-07-30 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Acute Coronary Syndrome; STEMI; Coronary Occlusion; Coronary Syndrome; NSTEMI; NSTEMI - Non-ST Segment Elevation MI
Keywords: Acute Coronary Syndrome; ECG; Artificial Intelligence; Occlusion Myocardial Infarction; Myocardial Infarction (MI)
MeSH Terms: conditions — Acute Coronary Syndrome; ST Elevation Myocardial Infarction; Coronary Occlusion; Angina, Unstable; Non-ST Elevated Myocardial Infarction; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
AI ECG TIMI is an investigator-initiated, international, and multicenter registry of acute coronary syndrome patients aimed to identify electrocardiographic findings detected by an AI model predicting coronary blood flow alteration. The aim of the study is to identify electrocardiographic findings detected by an automated artificial intelligence (AI) model that can predict coronary blood flow alteration as assessed by the TIMI grade flow at the very moment of the invasive coronary angiography in patients with acute coronary syndromes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute coronary syndromes undergoing invasive coronary angiography as clinically indicated.
* Availability of a standard 12-lead ECG performed at invasive coronary angiogram before percutaneous coronary intervention (maximum within 15 min before vascular access).
* Age ≥18 years.

Exclusion Criteria:

* Individuals presenting for a non-emergent (elective) cardiac catheterization.
* Individuals presenting with chronic coronary syndrome (CCS) or stable angina symptoms.
* Individuals without symptoms suspicious for acute coronary syndromes.
* Individuals with contraindications for cardiac catheterization.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (18 or older) with acute coronary syndrome undergoing clinically indicated invasive coronary angiography, with a standard 12-lead ECG performed at invasive coronary angiogram before percutaneous coronary intervention (maximum within 15 min before vascular access)
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of the AI-ECG TIMI AI Model | Index hospitalization (assessed up to 5 days)
  The primary endpoint is the AI-ECG TIMI model's ability to identify patients with actively occluded (TIMI 0-1) at the time of invasive coronary angiography using only single-standard 12-lead ECGs assessed by accuracy, sensitivity, specificity, positive, negative predictive values and F1 scores.

SECONDARY OUTCOMES:
Subgroup Performance | Index hospitalization (assessed up to 5 days)
  AI-ECG TIMI AI Model's performance across subgroups
  1. Demographic
  2. Risk factors & co-morbidities
  3. Electrocardiographic
  4. Culprit artery territory
Correlate established definitions of occlusion myocardial infarction (OMI) to myocardial perfusion status | Index hospitalization (assessed up to 5 days)
  2. OMI definitions using routine angiographic and laboratory parameters will be correlated to abnormal myocardial perfusion using correlation coefficients.
ECG prediction of mechanical reperfusion | Index hospitalization (assessed up to 5 days)
  a. Correlation of AI-ECG TIMI model's raw numeric predictions (between 0 and 1) with myocardial perfusion grading post PCI.
Assessment of expert ECG interpretation blinded to all clinical information | Index hospitalization (assessed up to 5 days)
  1. Accuracy, sensitivity, specificity, positive and negative predictive value of expert interpretation of active OMI, reperfused OMI and entirety of OMI
  2. Inter-rater variability of expert interpretation of active OMI, reperfused OMI and entirety of OMI.
STEMI-equivalent ECG patterns | Index hospitalization (assessed up to 5 days)
  a. Prevalence of STEMI equivalent ECG patterns and their correlation to TIMI flow grade at angiography.
Subgroup analysis of NSTEMI-OMI patients | Index hospitalization (assessed up to 5 days)
  9. NSTEMI-OMI stratified according to immediate (<2h) vs. SoC (>2h) invasive management, median: i. Peak troponin (maximum rise before fall) ii. Median LVEF at discharge iii. Length of hospital stay iv. Length of cardiac care unit (CCU) or intensive care unit (ICU) stay v. Presence of life-threatening arrhythmias

CONTACTS AND LOCATIONS:
Overall Officials: Robert Herman, MD, PhD, Principal Investigator — Powerful Medical; Emanuele Barbato, MD, PhD, Study Chair — University of Roma La Sapienza; Jozef Bartunek, MD, PhD, Study Chair — Azorg Hospital, Aalst
Locations (9):
- Austria (3):
  - LKH Hochsteiermark, Standort Bruck, Bruck an der Mur
  - LKH II Standort West, Graz
  - Medical University of Graz, Graz
- Belgium (3):
  - OLV Aalst, Aalst
  - AZ Sint Jan, Bruges
  - Jessa Ziekenhuis, Hasselt
- Italy (3):
  - University Hospital D'Annunzio Chieti, Chieti
  - San Pietro Hospital, Rome
  - Sant´Andrea Hospital, Rome

IPD SHARING:
Plan to Share IPD: No